CLINICAL TRIAL: NCT00479986
Title: Effects of Pioglitazone in Patients With Type 2 Diabetes Mellitus and Coronary Heart Disease at High Risk for Vascular Complications : A Placebo-Controlled Study
Brief Title: Effects of Pioglitazone in Type 2 Diabetes Mellitus and Coronary Heart Disease
Acronym: PIOcard
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: IKFE Institute for Clinical Research and Development (Other)
Collaborators: Takeda (Industry); Johannes Gutenberg University Mainz (Other); Heidelberg University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ATS-K-016
Record Dates: First submitted 2007-05-29; First posted 2007-05-30 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2007-05

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease
Keywords: diabetes mellitus; monocyte activation; cardiovascular risk
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pioglitazone (Experimental)
  Interventions: Drug: pioglitazone
- placebo (Active Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pioglitazone
  Arms: Pioglitazone
Drug: placebo
  Arms: placebo

SUMMARY:
The goal of the study is to investigate the impact of a 4 week treatment with pioglitazone (in comparison to placebo) on biomarkers for atherosclerosis and cardiovascular risk, as well as the degree of activation of the immune system, when given on top of an anti-diabetic treatment (metformin and/or sulfonylurea drugs) that has already resulted in good glycemic control.

DETAILED DESCRIPTION:
PPARgamma activation by pioglitazone has shown to be associated with an improvement of cardiovascular risk when measured with clinical (assessement of intima-media-thickness) or biochemical (hsCRP, MMP-9 etc.) markers. Well controlled patients (HbA1c < 8.0 %) will receive either pioglitazone or placebo (randomised, double-blind) for 4 weeks. Blood will be drawn to investigate the change in cardiovascular or metabolic markers and mRNA will be isolated from circulating mononuclear cells to investiagte the degree of activation of the immune system, which is another measure for the risk of atherosclerosis development.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetes mellitus
* stable oral treatment with metfromin and/or sulfonylurea
* age 20 - 80 years
* angiographically confirmed atherosclerosis or hsCRP > 1 mg/l

Exclusion Criteria:

* type 1 diabetes
* HbA1c > 8.5 %
* severe disease
* acute coronary syndrome
* contraindications to pioglitazone (heart failure etc.)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2005-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Short-term effect of Pioglitazone on Markers of vascular risk (MMP-9, hsCRP, monocyte activation) | 4 weeks

SECONDARY OUTCOMES:
Safety | 4 weeks
Metabolic control (HbA1c, Glucose) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Forst, MD, Principal Investigator — IKFE - Institute for Clinical Research and Development, Mainz; Andreas Pfützner, MD, PhD, Study Director — IKFE - Institute for Clinical Research and Development, Mainz
Locations (2):
- Germany (2):
  - Dr. Michael Morcos, Heidelberg
  - IKFE, Mainz